CLINICAL TRIAL: NCT03367715
Title: A Phase II, Open-label, Single Arm Trial of Nivolumab, Ipilimumab, and Short-course Radiotherapy in Adults With Newly Diagnosed, MGMT Unmethylated Glioblastoma
Brief Title: Nivolumab, Ipilimumab, and Short-course Radiotherapy in Adults With Newly Diagnosed, MGMT Unmethylated Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00218
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: MGMT-unmethylated Glioblastoma (GBM); GBM
MeSH Terms: interventions — Nivolumab; Ipilimumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab + Ipilimumab + Short-course radiation therapy (Experimental): within 6 weeks of the first diagnostic surgery for glioblastoma, all subjects will initiate study treatment on Day 1
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Radiation: Radiation Therapy (RT)

INTERVENTIONS:
Drug: Nivolumab — study treatment on Day 1 with one dose of nivolumab 3 mg/kg
Drug: Ipilimumab — study treatment on Day 1 with one dose of ipilimumab 1mg/kg
Radiation: Radiation Therapy (RT) — total dose of 30 Gy, given in 5 consecutive fractions of 6 Gy each fraction.

SUMMARY:
This is a single arm, open-label, phase II trial of nivolumab, ipilimumab and short-course radiation therapy in adult patients with newly diagnosed, MGMT unmethylated GBM with the primary objective of determining the overall survival at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 years.
* Histopathological evidence of glioblastoma or gliosarcoma, WHO grade IV.
* Tumor MGMT promoter DNA not methylated (i.e., unmethylated) by central testing.
* Maximal tumor diameter (including residual tumor and resection cavity if subjects had tumor resection rather than only stereotactic biopsy) of 6.6 cm or less. Maximal tumor size allowed is derived from an estimated maximal radiotherapy planning target volume (PTV) of 150 cm3.
* Subjects must not have received any prior standard or investigational anti-tumor therapy other than surgery and must not intend to receive any standard or investigational anti-tumor therapy other than the study regimen.
* Karnofsky performance status (Appendix 2) of ≥60.
* Availability of a paraffin-embedded or frozen tumor-tissue block with a minimum of 1 cm2 of tumor surface area, or 20 unstained slides from the glioblastoma tissue specimen if a tumor block cannot be submitted.
* Subjects must start study agent within 6 weeks from the first diagnostic surgery for glioblastoma.
* An interval of at least 2 weeks for surgical resection and 1 week for stereotactic biopsy from the start of study treatment.
* A contrast-enhanced MRI must be obtained within 7 days of the first dose of study treatment.
* Adequate hematologic, hepatic, and renal function defined by

  * White blood cell count ≥ 2.0 x 109/L
  * Absolute neutrophil count ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Hemoglobin > 9 g/dL
  * Serum creatinine ≤1.5 x upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 40 mL/min according to the Cockcroft-Gault formula or local institutional standard method
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN
  * Total bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* Women of child-bearing potential (WOCBP) and men able to father a child must agree to use highly effective contraception (any contraceptive method with a failure rate of less than 1% per year) while on study drug and for 23 weeks (for women) or 31 weeks (for men) after the last dose of study drug.

  1. WOCBP must have a negative serum or urine pregnancy test within 24 hours of initiation of study drug.
  2. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL to be defined as post-menopausal.
  3. WOCBP receiving nivolumab will be instructed to adhere to contraception for a period of 23 weeks after the last dose of investigational product. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. These durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days and men who are sexually active with WOCBP use contraception for 5 half-lives plus 90 days.
  4. Highly effective contraceptive measures include: stable use of oral contraceptives such as combined estrogen and progestogen and progestogen only hormonal contraception or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; intrauterine hormone-releasing system (IUS); bilateral tubal ligation; vasectomy and sexual abstinence.
  5. Contraception is not required for men with documented vasectomy.
  6. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.
  7. Women must not be breastfeeding.
* Willing to and capable of providing written informed consent prior to any study related procedures.
* Ability and willingness to comply with all study requirements, including scheduled visits, treatment plans, laboratory tests, and other study-related procedures.

Exclusion Criteria:

* Prior use of any standard or investigational anti-tumor therapy other than surgery
* Planned participation in another study of an investigational agent or investigational device or planned use of any other agent or therapeutic device intended for therapy of glioma.
* Prior systemic treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
* Primary brainstem or spinal cord tumor.
* Diffuse leptomeningeal gliomatosis.
* Known mutation of the IDH1 or IDH2 genes in the tumor, since glioblastomas with these mutations have different biology and are associated with improved prognosis.
* Systemic treatment with either immunosuppressive doses of corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration.

  1. Subjects on a standard high-dose steroid taper after craniotomy or stereotactic biopsy may have received a higher dose of corticosteroids within 14 days of registration, however must be at a dose < 10 mg daily prednisone or bioequivalent per day within 5 days prior to initiation of study drug.
  2. Administration of steroids through a route known to result in a minimal systemic exposure [i.e., intranasal, intraocular, inhaled, topical, or local injection (e.g., intra-articular injection) corticosteroids (<5% of body surface area)] are permitted in the absence of active autoimmune disease.
  3. Subjects requiring adrenal replacement with corticosteroids are eligible if the steroids are at doses ≤ 10 mg prednisone or bioequivalent per day in the absence of active autoimmune disease.
  4. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) are allowed.
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. The following conditions are not exclusions (subjects with the following conditions are permitted):

  a.Patients with diabetes type I, vitiligo, residual hypo- or hyperthyroidism due to autoimmune condition only requiring hormone replacement, or psoriasis not requiring systemic immunosuppressive treatment, or autoimmune conditions not expected to recur in the absence of an external trigger.
* Prior organ transplantation, including allogeneic stem cell transplantation.
* Known history of, or any evidence of active, non-infectious pneumonitis within the last 5 years.
* Known severe (NCI-CTCAE v4.03 Grade 3 or 4) infusion-related allergy or acute hypersensitivity reaction attributed to any monoclonal antibody, any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).
* Unable tolerate an MRI, or have a contraindication to MRI.
* Active infection requiring systemic therapy.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
* Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus (HCV antibody) indicating acute or chronic infection.
* Vaccination within 4 weeks of the first dose of study drug and while on trials is prohibited except for administration of inactivated vaccines. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Patients with another active cancer [excluding basal cell carcinoma, cervical carcinoma in situ or melanoma in situ]. Prior history of other cancer is allowed, as long as there was no active disease within the prior 2 years.
* All other unstable, severe, or chronic medical or psychiatric conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis, recent (within the past year) or active suicidal ideation or behavior, known alcohol or drug abuse, or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2022-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Chi, MD, Principal Investigator — NYU Langone Health; Sylvia Kurz, MD, Principal Investigator — NYU Langone Health; Erik Sulman, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab + Ipilimumab + Short-course Radiation Therapy
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab + Ipilimumab + Short-course Radiation Therapy
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 56 [46 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: 1-year Overall Survival (OS)
Description: Survival rate is defined as the percentage of participants who survived at 1 year (from either the date of diagnosis or the start of treatment for a disease)
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab + Ipilimumab + Short-course Radiation Therapy
Number analyzed (Participants) | 10
percentage of participants | 80

2. Secondary Outcome: Median Overall Survival (OS)
Description: Median survival rate of evaluable participants will be reported in months of survival
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Nivolumab + Ipilimumab + Short-course Radiation Therapy
Number analyzed (Participants) | 10
months | 16.85 [4.49 to 32.89]

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: The length of time during and after the treatment that a patient lives with the disease but it does not get worse.
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Nivolumab + Ipilimumab + Short-course Radiation Therapy
Number analyzed (Participants) | 10
months | 5.92 [1.48 to 13.93]

ADVERSE EVENTS:
Time Frame: 3 years
Description: Regular investigator assessment
Arm/Group | Nivolumab + Ipilimumab + Short-course Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 9/10
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab + Short-course Radiation Therapy (N=10)
Alanine Aminotransferase Increased (Investigations) | 6
Aspartate Aminotransferase Increased (Investigations) | 4
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab + Short-course Radiation Therapy (N=10)
Abdominal Pain (Gastrointestinal disorders) | 1
Agitation (Psychiatric disorders) | 1
Alkaline phosphatase increased (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 5
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Bruising (Injection Site) (Injury, poisoning and procedural complications) | 1
Central Nervous System Necrosis (Nervous system disorders) | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 2
Confusion (Psychiatric disorders) | 3
Conjunctivitis (Eye disorders) | 1
Creatinine Increased (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Dry eye (Eye disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Eye disorder, other; Diplopia (Eye disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
Insomnia (Psychiatric disorders) | 2
Lipase increased (Investigations) | 2
Localized Edema (General disorders) | 1
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 7
Lymphocyte count increased (Blood and lymphatic system disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oculomotor nerve disorder (Eye disorders) | 1
Pain (General disorders) | 1
Papulopustular Rash (Skin and subcutaneous tissue disorders) | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Platelet Count Decreased (Blood and lymphatic system disorders) | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pyramidal Tract Syndrome (Nervous system disorders) | 2
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 5
Restlessness (Psychiatric disorders) | 1
Serum Amylase Increased (Investigations) | 3
Sinus Bradycardia (Cardiac disorders) | 1
Skin + Subcutaneous tissue disorder (foot ulcer) (Skin and subcutaneous tissue disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary urgency (Renal and urinary disorders) | 1
Watering Eyes (Eye disorders) | 1
Weight Loss (Investigations) | 1
White Blood Cell Decreased (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT03367715/Prot_SAP_000.pdf